CLINICAL TRIAL: NCT06801756
Title: Description of Pregnancies and Their Impact on the Craniopharyngioma
Brief Title: Craniopharyngioma and Pregnancies
Acronym: CRANIOGESTE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241441
Record Dates: First submitted 2024-12-24; First posted 2025-01-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Craniopharyngioma
Keywords: pregnancy
MeSH Terms: conditions — Craniopharyngioma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The patients will respond to a questionnaire about their parental project, the occurence or not of complications during the pregnancy, and the impact of pregnancy on craniopharyngioma.

SUMMARY:
Craniopharyngiomas (CP) are rare hypothalamic-pituitary tumors found in young children, adolescents and adults. The management of PC remains complex, as their aggressive nature, invasive behavior and propensity to recur require sequential and balanced therapeutic attitudes, as well as follow-up in an expert center. Although patient survival rates are high, the consequences of the tumor and its treatment can lead to serious comorbidities and impaired quality of life, particularly in patients whose tumors extend to the hypothalamus. There is very little literature describing the outcome of pregnancy in craniopharyngioma patients and its impact on the craniopharyngioma. The largest study describes 6 women, mean age 24, who had a craniopharyngioma in childhood. Half of them had induced pregnancies; there is a succinct description of pregnancy complications and outcomes, as well as tumor progression.

In the endocrinology department of Pitié Salpêtrière hospital, the investigators regularly follow over a hundred patients of all ages who have presented with a craniopharyngioma in childhood or adulthood. They are also unique in having a medically assisted reproduction unit, which helps couples to realize their parental project. This dual specialization will enable to describe pregnancies and their impact on the behavior of craniopharyngiomas.

DETAILED DESCRIPTION:
Craniopharyngiomas are benign, slow-growing epithelial tumors that develop from the pituitary stem or pituitary gland in the sellar and/or parasellar region. They account for 2-4% of intracranial tumours and 5.6-15% of childhood tumours. The age distribution at diagnosis of these tumors is bimodal, with a first peak of incidence in children aged 5 to 14, and a second peak in adults aged 50 to 74. Despite the benign nature of these lesions, the quality of life of affected patients is most often impaired, due to endocrine (panhypopituitarism, hypothalamic obesity), visual and neuro-intellectual sequelae associated with the tumor itself and/or its treatment, as well as a high rate of local recurrence.

Treatment is mainly surgical, with the aim of removing as much of the tumour as possible and reducing the rate of local recurrence. However, this procedure has a high morbidity and mortality rate, without preventing a significant risk of recurrence (up to 62% at 10 years). Treatment is often complemented by radiotherapy or proton therapy to improve tumor control. Craniopharyngioma patients have an overall mortality rate 3 to 5 times higher than that observed in the general population. Increased morbidity is also observed in relation to hypopituitarism, hypothalamic lesions, visual and neurocognitive deficits, reduced quality of life and the development of cardiovascular risk factors.

The literature describing pregnancy in women with craniopharyngioma and the impact on the tumor is almost non-existent. A case report published in 2002 relates the story of a patient whose craniopharyngioma was discovered following visual disturbances and operated on at the age of 8; she presented with secondary panhypopituitarism, other complications are not mentioned. She became pregnant at the age of 34 after 8 cycles of gonadotropin stimulation. The pregnancy was uneventful and she delivered at term after spontaneous labor a eutrophic daughter weighing 3,450 g. She did not lactate. During pregnancy, it was necessary to increase the doses of L-thyroxine, hydrocortisone and desmopressin, which were resumed at the usual doses 3 weeks after delivery. No mention was made of changes in tumour volume, visual disturbances, neurocognitive disorders or weight gain during pregnancy. The largest study described 6 women, mean age 24, who had had a craniopharyngioma in childhood. Four of them had at least one pituitary deficiency, half of them had had induced pregnancies; there appeared to be no obstetric complications, no description was made of tumor evolution, hormone substitutions, weight.

The aim of this study is to carry out a monocentric study on patients followed in the endocrinology and reproductive medicine department of the Pitié-Salpêtrière hospital.

This department is the constituent center of the CRESCENDO CRMR, which includes craniopharyngiomas, and one of the reference endocrinology departments for craniopharyngiomas in Ile-de-France, so it has the expertise and one of the largest populations of patients with this rare pathology in the region.

The cohort is the result of two main recruitments:

* Craniopharyngiomas revealed in childhood: by pediatric endocrinology departments as part of the child-adult transition.
* Craniopharyngiomas diagnosed in adulthood: by the neurosurgery department of the Pitié-Salpêtrière hospital and by our private correspondents.

The literature on pregnancy in women with craniopharyngiomas is almost non-existent. The investigators would first like to know the proportion of women followed in the department who had a parental project, and whether the pregnancies were obtained naturally or through the use of antiretroviral treatment. They will describe the occurrence or non-occurrence of complications during pregnancy, the outcome of pregnancies and the impact of pregnancy on craniopharyngioma. To do this, the patients will be asked to fill in questionnaires relating mainly to their pregnancy, and the informations will be supplemented from medical records.

The investigators plan to carry out this work over a period of one year. They consider this period sufficient to mail the letter of information and non-opposition to the 100 patients eligible for this work.

Patients who do not object to their participation will then be contacted by telephone to complete a questionnaire. Each patient's participation will therefore last around thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years old
* Patients with or having had a craniopharyngioma
* Patients informed and not opposed to participation in research

Exclusion Criteria:

* Patients who don't speak french
* Patients without medical care insurance
* Patients under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female will be included
Study Population: Women with or having had a craniopharyngioma followed in the Endocrinology and Reproductive Medicine department at Pitié Salpêtrière, Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Describe how pregnancies are obtained: spontaneous or induced (and by which assisted reproduction technique). | 12 months
  Information on how the pregnancy was obtained will be collected from the medical record and will be completed on the day of inclusion by a telephone questionnaire with the patient.

SECONDARY OUTCOMES:
Describe the existence of a parental project among the women in the cohort | 12 months
  Information on the existence of a parental project will be completed on the day of inclusion by a telephone questionnaire with the patient.
Describe obstetric outcomes | 12 months
  Describe obstetric outcomes from the informations obtained during the telephone questionnaire, and pregnancy/childbirth reports.
Describe hormonal replacement adaptations. | 12 months
  From the prescriptions mentioned in the medical reports.
Describe the evolution of tumor volume during pregnancy or postpartum | 12 months
  From the informations mentioned in the medical reports.
Describe the visual impact if any | 12 months
  From ophthalmological reports
Describe the neurocognitive disorders if any | 12 months
  From neurological reports
Describe changes in weight during pregnancy | 12 months
  From the informations obtained during the telephone questionnaire, and pregnancy/childbirth reports (in kilograms).

CONTACTS AND LOCATIONS:
Overall Officials: Anne BACHELOT, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal